CLINICAL TRIAL: NCT06752317
Title: Effect of Preoperative Intrathecal Dexamethasone Versus Dexmedetomidine on Paralytic Ileus After Major Abdominal Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Hamed, resident doctor at Assiut University hospital, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dexamethasone vsdexmedetomidin
Record Dates: First submitted 2024-12-22; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Paralytic Ileus
Keywords: major abdominal surgery
MeSH Terms: conditions — Intestinal Pseudo-Obstruction | interventions — Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexamethasone group (Experimental): patients will receive intrathecal dexamethasone 8 mg in 3 ml volume.
  Interventions: Drug: Dexamethasone
- Dexmedetomidine group (Experimental): patients will receive intrathecal dexmedetomidine 0.5 µg/kg in 3 ml volume.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexamethasone — patients will receive intrathecal dexamethasone 8 mg in 3 ml volume.
  Arms: Dexamethasone group
Drug: Dexmedetomidine — patients will receive intrathecal dexmedetomidine 0.5 µg/kg in 3 ml volume.
  Arms: Dexmedetomidine group

SUMMARY:
Postoperative Ileus (POI) is considered as intolerance of oral intake due to disruption of the normal coordinated propulsive motor activity of the gastrointestinal (GI) tract following abdominal or non-abdominal surgery.

Dexamethasone & Dexmedetomidine have been reported to attenuate the incidence of paralytic ileus after abdominal surgeries.

Previous study has shown that a single dose of DM before induction of anesthesia may be beneficial to reduce ileus for IBD by alleviating the postoperative systemic inflammatory response.

Perioperative dexmedetomidine in major abdominal surgeries significantly decreased the time to flatus, defecation, and resuming normal diet, shortened length of stay, and improved haemodynamic stability.

The aim of this study is to compare the effect of preoperative intrathecal dexamethasone versus dexmedetomidine on paralytic ileus after major abdominal surgery.

DETAILED DESCRIPTION:
Postoperative Ileus (POI) is considered as intolerance of oral intake due to disruption of the normal coordinated propulsive motor activity of the gastrointestinal (GI) tract following abdominal or non-abdominal surgery.

Dexamethasone & Dexmedetomidine have been reported to attenuate the incidence of paralytic ileus after abdominal surgeries.

Previous study has shown that a single dose of DM before induction of anesthesia may be beneficial to reduce ileus for IBD by alleviating the postoperative systemic inflammatory response.

Perioperative dexmedetomidine in major abdominal surgeries significantly decreased the time to flatus, defecation, and resuming normal diet, shortened length of stay, and improved haemodynamic stability.

ELIGIBILITY:
Inclusion Criteria:

* • Age: 18-60 years.

  * Sex: both males and females.
  * ASA physical status: I and II.
  * Operation: Open major abdominal surgery.
  * The surgery has to involve gastrointestinal resection and/or anastomosis.

Exclusion Criteria:

* • History of abnormal bowl habit or bowel obstruction

  * Allergy to dexamethasone or dexmedetomidine
  * Electrolyte disturbance
  * Patient who receive any drugs known to influence gastrointestinal motility.
  * Mental disorders or inability to cooperate
  * Morbid obesity (BMI > 40), pregnancy, lactation
  * Diabetes
  * After neoadjuvant chemotherapy.
  * History of use of any steroids within the last 3 months
  * Previous abdominal surgery, herniorrhaphy or unplanned secondary surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative vomiting | 24 hours
  number of participants who had experienced vomiting on day 1.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abernethy EK, Aly EH. Postoperative Ileus after Minimally Invasive Colorectal Surgery: A Summary of Current Strategies for Prevention and Management. Dig Surg. 2024;41(2):79-91. doi: 10.1159/000537805. Epub 2024 Feb 15. PMID 38359801
- [Background] Chen Y, Dong C, Lian G, Li D, Yin Y, Yu W, Du C, Liu C, Li L, Tian F, Jing C. Dexamethasone on postoperative gastrointestinal motility: A placebo-controlled, double-blinded, randomized controlled trial. J Gastroenterol Hepatol. 2020 Sep;35(9):1549-1554. doi: 10.1111/jgh.15020. Epub 2020 Mar 5. PMID 32103514
- [Background] Zhang T, Xu Y, Yao Y, Jin L, Liu H, Zhou Y, Gu L, Ji Q, Zhu W, Gong J. Randomized Controlled Trial: Perioperative Dexamethasone Reduces Excessive Postoperative Inflammatory Response and Ileus After Surgery for Inflammatory Bowel Disease. Inflamm Bowel Dis. 2021 Oct 20;27(11):1756-1765. doi: 10.1093/ibd/izab065. PMID 33749741
- [Background] Lee MJ, Vaughan-Shaw P, Vimalachandran D; ACPGBI GI Recovery Group. A systematic review and meta-analysis of baseline risk factors for the development of postoperative ileus in patients undergoing gastrointestinal surgery. Ann R Coll Surg Engl. 2020 Mar;102(3):194-203. doi: 10.1308/rcsann.2019.0158. Epub 2019 Dec 20. PMID 31858809